CLINICAL TRIAL: NCT06732778
Title: Effectiveness of Pain Neuroscience Education in Women With Menstrual Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, osman coban, Asst. Professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Uskudaruniversity5
Record Dates: First submitted 2024-12-09; First posted 2024-12-13 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Pain Management; Dysmenorrhea (Disorder)
Keywords: dysmenorrhea; pain; quality of life; pain neuroscience education
MeSH Terms: conditions — Agnosia; Dysmenorrhea; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: randomized controlled Trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain neuroscience education group (PNE) (Experimental): The cases in this group will be given online PNE training one week before menstruation.
  Interventions: Other: Pain Neuroscience Education (PNE)
- Control Group (CG) (Other): No training or application will be given to the control group
  Interventions: Other: Control Group (CG)

INTERVENTIONS:
Other: Pain Neuroscience Education (PNE) — PNE was planned online for clients 1 week before menstruation in the form of speaking sessions in a presentation format. The training will be conveyed in relation to pain during menstruation. Visual aids, examples and metaphors will be used to improve patient understanding in the training. Ankle sprain picture, speeding bus picture, action potential picture, picture showing membrane resting potential, rusty nail picture, whole body nervous system picture, neuromatrix picture, lion and lion cub picture that helps explain stress responses, curious neighbors picture etc. will be used. The training session is planned to last between 2 and 4 hours.
  The distribution of pain neuroscience training topics will be implemented in the order given below, with 10 main headings.
  * Pain and the Biopsychosocial Model
  * Injury and pain are not equivalent, pain is a brain output rather than an input
  * Action potential, normal electrical activity of nerves and conduction
  * Biological process of ion chann
  Arms: Pain neuroscience education group (PNE)
Other: Control Group (CG) — The control group will not receive any training or practice.
  Arms: Control Group (CG)

SUMMARY:
Menstruation is the bleeding that starts with menarche and continues until menopause, along with hormonal changes in women of reproductive age, and is shed as the endometrium matures and is shed. Menstruation, which covers 30-35 years of a woman's life and occurs regularly every month, is a physiological process. Menstrual cycle problems are a condition that affects health and society all over the world and causes treatment to be sought. It is one of the most common menstrual cycle problems.

Dysmenorrhea is used synonymously with menstrual pain in clinics and practice. It is stated that approximately 40-50% of women experience dysmenorrhea and that it is more common in adolescents. Dysmenorrhea is a symptom that causes changes in women's physical activities and social roles, leading to a decrease in their quality of life. Dysmenorrhea usually manifests itself with symptoms such as pain and cramps in the back and lower abdomen, as well as nausea, vomiting, fatigue, irritability, appetite changes, diarrhea, and headache.

According to the literature, among the choices of women to cope with dysmenorrhea, manipulative and body-based practices (massage, relaxation exercises, acupuncture, aromatherapy, hot-cold applications, etc.), mind-body-based practices (meditation, yoga, hypnotherapy, hypnosis, music therapy, etc.), vitamin-mineral supplements and herbal therapies (vitamins B and E, magnesium, zinc, fennel/rose tea, black cohosh, etc.) and exercise programs are seen to be effective.

DETAILED DESCRIPTION:
The first concepts of pain neuroscience education emerged in 2002 in a randomized controlled trial conducted by Lorimer Moseley for patients with low back pain. PNE has been given various names, including but not limited to pain biology education, pain neurophysiology education, neuroscientific pain education, and neuroscience education. In general, PNE is an educational intervention that aims to explain to the patient the neurophysiology of pain, nervous system sensitivity, nervous system plasticity, and psychosocial factors that contribute to the experience of persistent pain. This is accomplished through a series of intertreatment educational modules spread over a term. The modules include exposure to visual aids, examples, and metaphors to enhance patient understanding. The duration and frequency of educational sessions are not uniform in the literature; they range from 30 minutes to 4 hours. Pain neuroscience education connects the pathoanatomical model of tissue damage with the neurophysiological and psychosocial factors inherent in the experience of persistent pain. The goal is to help patients reconceptualize their pain experience by providing educational content that can reduce focus on anatomic damage, decrease fear avoidance, reduce kinesiophobia, and improve self-efficacy. The exact dosage, frequency, and content of a PNE intervention vary.

There are studies in the literature examining the effectiveness of PNE in chronic low back pain, chronic whiplash injury, chronic fatigue syndrome, and the postoperative and preoperative periods of lumbar surgery. No study was found using the pain neuroscience education method in clients with menstrual period pain.

The aim of this study was to investigate the effectiveness of pain neuroscience education on pain and quality of life in women with menstrual period pain.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age,
* Not having a previous pregnancy,
* Not having a history of pelvic infections
* Not using hormonal contraception and intrauterine devices,
* Having a menstrual period of 3-8 days and a menstrual cycle interval of 21-35 days,
* Being willing to participate in the study.

Exclusion Criteria:

* Being under 18 years of age,
* Having a previous pregnancy,
* Having a history of pelvic infections
* Using hormonal contraception and intrauterine devices,
* Not having a menstrual period of 3-8 days and a menstrual cycle interval of 21-35 days,
* Not being willing to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Menstruation
Enrollment: 74 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Scale for Assessing the Impact of Dysmenorrhea on Daily Life (SAIDDL) | 4 weeks
  The Scale for Assessing the Impact of Dysmenorrhea on Daily Life was prepared to determine and compare the extent to which daily life is affected by the pain experienced during menstruation. On the 3rd day of each menstrual period, the degree to which daily life is affected is marked on the horizontal line with the numerical values between 0 and 10. A score of 0 on the scale indicates that daily life is "not affected at all" by dysmenorrhea, while a score of 10 indicates that it is "completely affected".

SECONDARY OUTCOMES:
Pain Beliefs Scale (BPS) | 4 weeks
  It was developed by Edwards and colleagues in 1992. It has an 8-item Organic Beliefs subtest (items 1, 2, 3, 5, 7, 8, 10, 11) and a 4-item Psychological Beliefs subtest (items 4, 6, 9, 12). When the scale is applied, the person is asked to mark the most appropriate option for themselves from 6 options ranging from "never" to "always". Scoring varies between 1 and 6 for each item. The total score for each subtest is calculated by adding the scores from the items in the relevant subtest and dividing them by the number of items in the relevant subtest, and three score types (organic beliefs subscale, psychological beliefs subscale, and total score) are obtained.
McGill Pain Scale Short Form (MSS-SF) | 4 weeks
  The McGill Pain Scale Short Form consists of three sections. Section One: This section contains 15 descriptive word groups. 11 of these evaluate the sensory and 4 evaluate the perceptual dimensions of pain. These descriptive words are rated on an intensity scale between 0 and 3 (0=none, 1=mild, 2=moderate, 3=extreme). In the first section of the scale, a total of 3 pain scores are obtained: sensory pain score, perceptual pain score, and total pain score. Section Two: The second section of the form contains five word groups ranging from "mild pain" to "unbearable pain" to determine the severity of the patient's pain. Section Three: In the third section, the patient's current pain intensity is evaluated using a visual comparison scale.

CONTACTS AND LOCATIONS:
Overall Officials: osman coban, Asst Prof., Study Director — Uskudar University; cigdem inkaya, PT, Principal Investigator — Uskudar University
Locations (1):
- Uskudar University, Faculty of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zimney K, Van Bogaert W, Louw A. The Biology of Chronic Pain and Its Implications for Pain Neuroscience Education: State of the Art. J Clin Med. 2023 Jun 21;12(13):4199. doi: 10.3390/jcm12134199. PMID 37445234
- [Result] O'Connor M, Sillevis R, Erickson MR. Pain Neuroscience Education Delivered by a Student Physical Therapist for a Patient with Persistent Musculoskeletal Pain. Am J Case Rep. 2021 Aug 16;22:e932212. doi: 10.12659/AJCR.932212. PMID 34398869
- [Result] Louw A, Farrell K, Choffin B, Foster B, Lunde G, Snodgrass M, Sweet R, Weitzel M, Wilder R, Puentedura EJ. Immediate effect of pain neuroscience education for recent onset low back pain: an exploratory single arm trial. J Man Manip Ther. 2019 Dec;27(5):267-276. doi: 10.1080/10669817.2019.1624006. Epub 2019 Jun 4. PMID 31161919
- [Result] Sillevis R, Trincado G, Shamus E. The immediate effect of a single session of pain neuroscience education on pain and the autonomic nervous system in subjects with persistent pain, a pilot study. PeerJ. 2021 May 31;9:e11543. doi: 10.7717/peerj.11543. eCollection 2021. PMID 34131526